CLINICAL TRIAL: NCT03070054
Title: LIA in Hip Arthroscopy Patients: An Extra-Capsular Approach
Brief Title: LIA in Hip Arthroscopy Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90371
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2020-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants, anesthesiologists and PACU nurses will be blinded to group assignment, however the surgeon administering the LIA will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): non-LIA group prior to surgery
- Treatment (Experimental): Extra-capsular local infiltration analgesic (LIA) administration of 20ml 0.25% bupivacaine-epinephrine
  Interventions: Drug: 20ml 0.25% bupivacaine-epinephrine

INTERVENTIONS:
Drug: 20ml 0.25% bupivacaine-epinephrine — Extra-capsular local infiltration analgesic (LIA) administration of 20ml 0.25% bupivacaine-epinephrine
  Other Names: Marcaine, Sensorcaine
  Arms: Treatment

SUMMARY:
The investigator's are conducting a randomized, blinded study to determine if the extra-capsular local infiltration analgesic (LIA) administration of 20ml 0.25% bupivacaine-epinephrine can improve the postoperative pain management of hip arthroscopy patients. Participants will be randomly assigned to the LIA group or non-LIA group prior to surgery. Participants, anesthesiologists and PACU nurses will be blinded to group assignment, however the surgeon administering the LIA will be unblinded.

DETAILED DESCRIPTION:
Hip arthroscopy is a growing field in orthopedic medicine that has gained momentum in recent years as a treatment for an array of hip pathologies including labral tears, chondral injuries, loose bodies, hip instability, femoroacetabular impingement, extraarticular lesions, synovial abnormalities, ruptured ligamentum teres, osteonecrosis, and mild-to-moderate osteoarthritis. With this increased rate of hip arthroscopy has come an interest in adequate postoperative pain management.

There are a number of strategies to improve post-operative orthopedic pain management. One common technique is the femoral block, during which a patient receives an ultrasound-guided injection of local analgesia administered in close proximity to the nerve. In the hip arthroscopy setting, postoperative femoral nerve blocks have been shown to significantly decrease pain, reduce opioid related symptoms like nausea, and have higher pain satisfaction scores than patients using only morphine. However, this option can be costly as it is a separate procedure billed by the anesthesiologist. Regional nerve blocks also carry the risk of residual parasthesia and permanent nerve damage, however rare.

One way to circumvent these limitations is through local infiltration analgesia (LIA), a technique that has been described for post-operative pain management in orthopedic modalities like total knee arthroscopy (TKA) and total hip arthroscopy (THA). Injection of analgesic directly to the surgical site can easily be incorporated as a brief step in the surgical procedure at a minimal cost to the patient. In THA and TKA, LIA has resulted in promising decreases in pain and opioid consumption. However, interpretation of these results in the context of hip arthroscopy has been confounded by the fundamental differences between THA/TKA and hip arthroscopy, the array of different strategies used in LIA (eg. continuous infiltration via a catheter vs. a single shot), and a lack of placebo or control group, and the specific location of injection.

In the setting of hip arthroscopy, a previous group tested intra-portal injections with mixed results. LIA targeting the highly innervated hip capsule, which is cut to access the joint during arthroscopy, may be more efficacious at limiting postoperative pain. LIA injection into the hip capsule can occur under direct visualization after capsular repair. To our knowledge, no studies have assessed the outcomes of this extracapsular LIA technique in the hip arthroscopy setting.

Documented risks involved with LIA are limited to the continuous infiltration via catheter. This approach has the risk of infection at the catheter site as well as cartilage damage. Our proposed technique avoids use of catheters and associated infection. The proposed single dose of 0.25% 20mL bupivacaine epinephrine a fraction of the dosages used in previous LIA studies to avoid chondral damage.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) patients who have elected for hip arthroscopy surgery.

Exclusion Criteria:

* Patients who are undergoing bilateral hip arthroscopy in a single surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
PACU pain scores | 1-day
  Patient-reported pain in the postoperative anesthesia care unit (PACU).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aoki, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No